CLINICAL TRIAL: NCT07287176
Title: Prospective Evaluation of the Pulse Biosciences nPulse™ Vybrance™ Percutaneous Electrode System in Symptomatic Benign Thyroid Nodules (PRECISE-BTN) Study
Brief Title: Prospective Evaluation of the Pulse Biosciences nPulse™ Vybrance™ Percutaneous Electrode System
Acronym: PRECISE-BTN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-TF-US-038
Record Dates: First submitted 2025-12-11; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Nodule; Thyroid Goiter; Ablation
Keywords: nsPFA; Pulsed Field Ablation
MeSH Terms: conditions — Thyroid Nodule; Goiter

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, single arm, non-randomized, feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- nPulse Vybrance Percutaneous Electrode System Treatment Arm (Experimental): Adult participants who are clinically symptomatic will receive ablation of the benign thyroid nodule using the nPulse Vybrance Percutaneous Electrode System.
  Interventions: Device: nPulse Vybrance Percutaneous Electrode System

INTERVENTIONS:
Device: nPulse Vybrance Percutaneous Electrode System — The nPulse Vybrance procedure will be performed under ultrasonographic guidance using a local anesthetic at the intended puncture site and all participants will receive general anesthesia in the operating room. The targeted thyroid nodule will be treated within a customized treatment level (DEFAULT) programmed on the Console. The Investigator will treat the entire nodule while protecting from ablation to any surrounding vital structures to prevent serious adverse events throughout the procedure. Any procedural adverse events will be documented, as applicable.

SUMMARY:
The primary objective of this study is to reproduce in a multi-center study results obtained during the feasibility First-In-Human (FIH) study with Prof. Stefano Spiezia, MD (Ospedale del Mare, Naples, Italy) and to monitor additional thyroid-related symptoms and impact of patients quality of life post-ablation using a validated QoL questionnaire.

DETAILED DESCRIPTION:
The study design is a prospective, non-randomized, clinical study using the Pulse Biosciences nPulse Vybrance Percutaneous Electrode (PE) System for the treatment of benign thyroid nodules (BTNs) using nanosecond Pulsed Field Ablation (PFA). All participants will receive at least one nsPFA treatment and may be eligible to receive a second treatment at the 6-month follow up visit per physician discretion. All participants will have regularly scheduled ultrasound assessments and administration of questionnaires (e.g., Thy-PRO39 and SF-12) at 1-month, 3 months, 6 months and 12 months post-nsPFA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to provide voluntary, written informed consent to participate in this study and from whom written informed consent has been obtained
* Participants must be willing and able to comply with study procedures including all follow-up visits
* Selected nodule is amenable to trans-isthmus approach
* Nodule is confirmed as benign based on results from one or more of the following diagnostic tests:

  1. (Bethesda II) on at least 2 ultrasound guided fine needle aspirations (FNA) or core needle biopsy (CNB);
  2. A single benign diagnosis of FNA or CNB when the nodule has benign ultrasound features [American College of Radiology (ACR) Thyroid Imaging Reporting & Data System [TI-RAD] TR 1-3, American Thyroid Association [ATA] very low suspicion];
  3. Candidate has a hyperfunctional nodule following 1 ultrasound guided FNA or CNB with or without molecular testing; or
  4. Benign (Bethesda III or IV) with two biopsies in addition to molecular testing confirming benign diagnosis
* Selected nodule is <80.0 ml
* Participant has normal vocal cord mobility by ultrasound evaluation
* Participant has presence of compression symptoms, cosmetic concerns or anxiety for which participant requests treatment of the benign thyroid nodule
* Participant has a solitary thyroid nodule or dominating nodule that is well-defined in multinodular goiter

Exclusion Criteria:

* Participant has an implantable electronic medical device. (i.e., pacemaker, implantable cardioverter defibrillator)
* Participant has cystic nodules (< 70% solid components)
* Participant has calcified nodules
* Participant is known to be immune compromised
* Participant had previous neck irradiation
* Participant has abnormal cervical lymph nodes present during screening visit examination
* Participant has history of familial thyroid cancer in more than two first-degree relatives
* Selected nodule previously treated with radiofrequency ablation or ethanol. This does not apply to nodules previously treated with nanosecond Pulsed Field Ablation (nsPFA)
* Participants currently suffering from a hematological disease or bleeding tendency
* Selected nodule likely to be in contact with the recurrent laryngeal nerve on ultrasound evaluation
* Participant has a history of uncontrolled cardiac arrhythmia, uncontrolled hypertension, chronic liver disease or chronic kidney disease (Stage 4-5), or recent history of myocardial infarction or structural heart disease as determined by the Investigator
* Participant has abnormal contralateral vocal cord function
* Anesthesia drug allergies
* Participant is pregnant at the time of screening or within 30 days prior to enrollment
* Participant has any condition or situation which, in the Investigator's opinion, puts the participant at significant risk, could confound the study results, or may interfere significantly with the participant's participation in the study
* Use of any investigational device or drug within 30 days prior to enrollment that may confound the results of this study

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Volume Reduction Ratio (VRR) | 6 months post-index procedure
  The percentage decrease of thyroid nodule volume measured by ultrasonography after treatment (ablation) using the nPulse Vybrance Percutaneous Electrode System

SECONDARY OUTCOMES:
Volume Reduction Ratio (VRR) Over Time | 1 month, 3 months, 6 months and 12 months post-nPulse Vybrance treatment
  The percentage decrease of thyroid nodule volume measured by ultrasonography after treatment (ablation) at various time points post-ablation using the nPulse Vybrance Percutaneous Electrode System
Recurrence Rate | 6 and 12 months post-nPulse Vybrance treatment
  The number of participants who experience nodule recurrence in same location of treatment post-nPulse Vybrance index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Tufano, MD, Principal Investigator — Sarasota Memorial Hospital
Locations (2):
- United States (2):
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No